CLINICAL TRIAL: NCT00004376
Title: Phase III Randomized, Double-Blind, Placebo-Controlled Study of Guanfacine for Tourette Syndrome and Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Yale University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11979; YALESM-7588
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-03

CONDITIONS: Tourette Syndrome
Keywords: Tourette syndrome; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Tourette Syndrome; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Guanfacine

INTERVENTIONS:
Drug: guanfacine

SUMMARY:
OBJECTIVES:

I. Evaluate the safety and efficacy of the alpha-2 adrenergic agonist guanfacine in children and adolescents with Tourette syndrome or other chronic tic disorder, and attention deficit hyperactivity disorder.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind study. Patients are stratified by pubertal status.

There is a 7- to 14-day washout with a placebo prior to treatment for all patients.

The first group receives oral guanfacine 3 times a day for 8 weeks. The dose is gradually increased to minimize sedation; by day 14, most patients are stabilized and the dose is then increased as clinically indicated and tolerated.

The second group receives a placebo 3 times a day for 8 weeks. Patients in either group may be treated with guanfacine for an additional 8 weeks.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Tourette syndrome or other chronic tic disorder meeting Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) criteria
* DSM-IV diagnosis of attention deficit hyperactivity disorder (ADHD) Clinician's Global Impression for ADHD greater than 4 Hyperactivity Index of Conners Parent or Teacher Questionnaire standard score 65 or higher (1.5 standard deviation units)

--Prior/Concurrent Therapy--

* At least 2 weeks since medication for tics, ADHD, or obsessive compulsive disorder (4 weeks since neuroleptics or fluoxetine)
* No failure on prior guanfacine

--Patient Characteristics--

* Hepatic: No liver failure
* Renal: No renal failure
* Cardiovascular: No hypertension No other heart disease
* Pulmonary: No pulmonary disease
* Other: No Intelligence Quotient below 80 No current DSM-IV diagnosis of the following: Major depression Bipolar disorder Pervasive developmental disorder Psychotic disorder No seizure disorder No other significant medical condition No pregnant women

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35
Dates: Start 1994-09; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Scahill, Study Chair — Yale University